CLINICAL TRIAL: NCT03703778
Title: Prospective Study of the Effect of Androgen Deprivation Therapy (ADT) in Male Patients Suffered Prostate Cancer in Asian Population
Brief Title: Real-life Evaluation of the Effect of ADT in Prostate Cancer Patients in Asia (READT Asia Study)
Acronym: READT
Status: Active, not recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, NG Chi Fai, Clinical Professor, Chinese University of Hong Kong
Other Study IDs: READT Asia
Record Dates: First submitted 2018-03-12; First posted 2018-10-12 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Androgen deprivation therapy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Leuprolide; luprolide acetate gel depot; acetyl-2-naphthylalanyl-3-chlorophenylalanyl-1-oxohexadecyl-seryl-4-aminophenylalanyl(hydroorotyl)-4-aminophenylalanyl(carbamoyl)-leucyl-ILys-prolyl-alaninamide

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- bilateral orchidectomy: Patients with advanced prostate cancer who receive surgical androgen deprivation therapy - bilateral orchidectomy
  Interventions: Procedure: Androgen deprivation therapy - bilateral orchidectomy
- GnRH agonist: Patients with advanced prostate cancer who receive medical androgen deprivation therapy - GnRH agonist
  Interventions: Drug: Androgen deprivation therapy - GnRH agonist
- GnRH antagonist: Patients with advanced prostate cancer who receive medical androgen deprivation therapy - GnRH antagonist
  Interventions: Drug: Androgen deprivation therapy - GnRH antagonist

INTERVENTIONS:
Procedure: Androgen deprivation therapy - bilateral orchidectomy — Androgen deprivation therapy (ADT) is a kind of hormone therapy for prostate cancer. The goal is to reduce levels of male hormones, called androgens, in the body, or to stop them from affecting prostate cancer cells. It can be surgical, i.e. bilateral orchidectomy, or medical, i.e. GnRH agonist or GnRH antagonist.
  Groups: bilateral orchidectomy
Drug: Androgen deprivation therapy - GnRH agonist — Androgen deprivation therapy (ADT) is a kind of hormone therapy for prostate cancer. The goal is to reduce levels of male hormones, called androgens, in the body, or to stop them from affecting prostate cancer cells. It can be surgical, i.e. bilateral orchidectomy, or medical, i.e. GnRH agonist or GnRH antagonist.
  Other Names: Enantone; Eligard
  Groups: GnRH agonist
Drug: Androgen deprivation therapy - GnRH antagonist — Androgen deprivation therapy (ADT) is a kind of hormone therapy for prostate cancer. The goal is to reduce levels of male hormones, called androgens, in the body, or to stop them from affecting prostate cancer cells. It can be surgical, i.e. bilateral orchidectomy, or medical, i.e. GnRH agonist or GnRH antagonist.
  Other Names: Degarelix
  Groups: GnRH antagonist

SUMMARY:
The prostate gland is a clinically important male accessory sex gland and vital for its production of semen. Prostate cancer (PCa) is now ranked 3th in annual incidence of male cancer and ranked 5th for cancer-related death in men in Hong Kong which accounts for about 10.9 deaths per 100,000 persons. Its incidence is rising rapidly, almost tripled in the past 10 years. Despite the improvement in awareness of the disease and also increasing use of serum prostate specific antigen, many patients still presented at a late stage that beyond cure by local therapy. Together with those patients suffered recurrent disease after local therapy, many PCa patients required the use of androgen deprivation therapy (ADT) for the control of disease.

However, unlike other malignancy, PCa is characterized by its slow progression nature and even for metastatic disease the 5-year survival is upto 20%. Therefore, while ADT can provide effective control of disease, there are increasing evidences suggesting that it can also result in many adverse effects in the patients, and these effects are particular important due to the long survival of these patients. From the western literature, the adverse effects can be quite diverse. Classical side effects after ADT include mood changes, hot flushes, change in cognitive function, loss of libido, erectile dysfunction, osteoporosis and pathological fracture, insulin resistance and increase in risk of cardiovascular related mortality.

Unfortunately information regarding the side effects of ADT in Asian population is scanty and inconclusive. Therefore, there is a need to have more information on the adverse effect profiles related to ADT in Asian population.

This is a multicentre, prospective, observational, non-interventional study to assess the clinical effectiveness, cardiometabolic and skeletal effects of the various type of ADT - bilateral orchidectomy, GnRH agonist, and GnRH antagonist - in men with advanced prostate cancer over a minimum of 1-year observation period.

DETAILED DESCRIPTION:
The prostate gland is a clinically important male accessory sex gland and vital for its production of semen. Prostate cancer (PCa) is now ranked 3th in annual incidence of male cancer and ranked 5th for cancer-related death in men in Hong Kong which accounts for about 10.9 deaths per 100,000 persons. Its incidence is rising rapidly, almost tripled in the past 10 years. As the elderly population continues to increase, the impact of PCa on the men's health and also the burden on health care system will continue to rise.

Despite the improvement in awareness of the disease and also increasing use of serum prostate specific antigen, many patients still presented at a late stage that beyond cure by local therapy. Together with those patients suffered recurrent disease after local therapy, many PCa patients required the use of androgen deprivation therapy (ADT) for the control of disease.

However, unlike other malignancy, PCa is characterized by its slow progression nature and even for metastatic disease the 5-year survival is upto 20%. Therefore, while ADT can provide effective control of disease, there are increasing evidences suggesting that it can also result in many adverse effects in the patients, and these effects are particular important due to the long survival of these patients. From the western literature, the adverse effects can be quite diverse. Classical side effects after ADT include mood changes, hot flushes, change in cognitive function, loss of libido, erectile dysfunction, osteoporosis and pathological fracture. Also there are more and more evidences showed ADT will also altered the metabolic and cardiovascular status of the patients and resulted in increase in insulin resistance and increase in risk of cardiovascular related mortality.

However, there is a lack of data concerning the association between ADT and various complications in the Asian population. Due to the genetic and physiological differences and the experience from studies on female menopause the cardiovascular risk profile may differ between different ethnicities. Reports from Japan suggested the effects of ADT in Japanese were different from Caucasian with better treatment efficacy and lower cardiovascular risk. However, reports from Hong Kong suggested the adverse effects of ADT in Chinese populations were quite similar to the reports in Western world. Moreover, due to the difference in social and cultural background in Asian countries, the usage of different modalities of ADT might be different in different areas, which might also affect the efficacy and outcomes in patients.

Therefore, investigator would like to perform a prospective study on the practice and effect of ADT in Asian population to try to clarify the effect of ADT in our regional population.

ELIGIBILITY:
Inclusion Criteria:

* All new, consecutive patients with histological proven prostate cancer or clinically diagnosed to have prostate cancer, who decided for ADT would be recruited for the study

Exclusion Criteria:

* Prior neoadjuvant or adjuvant hormone therapy within 1 year before
* Refuse or unable to give written informed consent
* Participation in an investigational program with interventions outside of routine clinical practice

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only male patients got prostate cancer
Study Population: Patients who come to our hospital urology specialist clinics and received androgen deprivative therapy will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2016-05-22 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients using surgical castration and medical castration in prostate cancer patients in Asia | 5 years
  The proportion of patients using surgical castration and medical castration in prostate cancer patients in Asia

SECONDARY OUTCOMES:
The incidence of cardiovascular complications in prostate cancer patients receiving androgen deprivation therapy | 5 years
  The incidence of cardiovascular complications, such as myocardial infarction, stroke, etc, in prostate cancer patients receiving different form of androgen deprivation therapy
The disease response in prostate cancer patients receiving different ADT | baseline, 6-month, 12 month, and then 6 monthly until 5 years
  To assess PSA progression in patients receiving different ADT

CONTACTS AND LOCATIONS:
Overall Officials: Chi Fai NG, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Shatin, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Beauchet O. Testosterone and cognitive function: current clinical evidence of a relationship. Eur J Endocrinol. 2006 Dec;155(6):773-81. doi: 10.1530/eje.1.02306. PMID 17132744
- [Background] Fang LC, Merrick GS, Wallner KE. Androgen deprivation therapy: a survival benefit or detriment in men with high-risk prostate cancer? Oncology (Williston Park). 2010 Aug;24(9):790-6, 798. PMID 20923031
- [Background] Lattouf JB, Saad F. Bone complications of androgen deprivation therapy: screening, prevention, and treatment. Curr Opin Urol. 2010 May;20(3):247-52. doi: 10.1097/MOU.0b013e32833835be. PMID 20224416
- [Background] Levine GN, D'Amico AV, Berger P, Clark PE, Eckel RH, Keating NL, Milani RV, Sagalowsky AI, Smith MR, Zakai N; American Heart Association Council on Clinical Cardiology and Council on Epidemiology and Prevention, the American Cancer Society, and the American Urological Association. Androgen-deprivation therapy in prostate cancer and cardiovascular risk: a science advisory from the American Heart Association, American Cancer Society, and American Urological Association: endorsed by the American Society for Radiation Oncology. Circulation. 2010 Feb 16;121(6):833-40. doi: 10.1161/CIRCULATIONAHA.109.192695. Epub 2010 Feb 1. No abstract available. PMID 20124128
- [Background] Namiki M, Ueno S, Kitagawa Y, Fukagai T, Akaza H. Effectiveness and adverse effects of hormonal therapy for prostate cancer: Japanese experience and perspective. Asian J Androl. 2012 May;14(3):451-7. doi: 10.1038/aja.2011.121. Epub 2012 Mar 26. PMID 22447200
- [Background] Rampp T, Tan L, Zhang L, Sun ZJ, Klose P, Musial F, Dobos GJ. Menopause in German and Chinese women--an analysis of symptoms, TCM-diagnosis and hormone status. Chin J Integr Med. 2008 Sep;14(3):194-6. doi: 10.1007/s11655-008-0194-1. Epub 2008 Oct 14. PMID 18853115
- [Background] Saylor PJ, Smith MR. Metabolic complications of androgen deprivation therapy for prostate cancer. J Urol. 2009 May;181(5):1998-2006; discussion 2007-8. doi: 10.1016/j.juro.2009.01.047. Epub 2009 Mar 14. PMID 19286225
- [Background] Smith MR. Treatment-related diabetes and cardiovascular disease in prostate cancer survivors. Ann Oncol. 2008 Sep;19 Suppl 7(Suppl 7):vii86-90. doi: 10.1093/annonc/mdn458. No abstract available. PMID 18790986
- [Background] Taylor LG, Canfield SE, Du XL. Review of major adverse effects of androgen-deprivation therapy in men with prostate cancer. Cancer. 2009 Jun 1;115(11):2388-99. doi: 10.1002/cncr.24283. PMID 19399748
- [Background] Teoh JY, Chiu PK, Chan SY, Poon DM, Cheung HY, Hou SS, Ng CF. Risk of ischemic stroke after androgen deprivation therapy for prostate cancer in the Chinese population living in Hong Kong. Jpn J Clin Oncol. 2015 May;45(5):483-7. doi: 10.1093/jjco/hyv025. Epub 2015 Feb 26. PMID 25724216
- [Background] Teoh JY, Chan SY, Chiu PK, Poon DM, Cheung HY, Hou SS, Ng CF. Risk of cardiovascular thrombotic events after surgical castration versus gonadotropin-releasing hormone agonists in Chinese men with prostate cancer. Asian J Androl. 2015 May-Jun;17(3):493-6. doi: 10.4103/1008-682X.143313. PMID 25578930
- [Background] Teoh JY, Chan SY, Chiu PK, Poon DM, Cheung HY, Hou SS, Ng CF. Risk of acute myocardial infarction after androgen-deprivation therapy for prostate cancer in a Chinese population. BJU Int. 2015 Sep;116(3):382-7. doi: 10.1111/bju.12967. Epub 2015 Mar 7. PMID 25327618
- [Background] Teoh JY, Chiu PK, Chan SY, Poon DM, Cheung HY, Hou SS, Ng CF. Risk of new-onset diabetes after androgen deprivation therapy for prostate cancer in the Asian population. J Diabetes. 2015 Sep;7(5):672-80. doi: 10.1111/1753-0407.12226. Epub 2014 Dec 22. PMID 25266491